CLINICAL TRIAL: NCT07086300
Title: Clinical Study of Electroacupuncture Combined With PD-1 Inhibitor Treatment for Elderly Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Electroacupuncture Combined With PD-1 Inhibitor for Elderly Patients With Advanced NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kong Fanming (Other)
Responsible Party: Sponsor-Investigator, Kong Fanming, Director of Oncology Department, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Organization: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TYLL2025[K]049
Record Dates: First submitted 2025-07-08; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Elderly Patients (>65 Years); Non-Small Cell Lung Cancer; PD-1 Inhibitors; Electroacupuncture
Keywords: electroacupuncture; Elderly patients; non-small cell lung cancer; Immunotherapy; immune checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Due to the specific nature of acupuncture clinical research, it is challenging to achieve double blinding of subjects and operators. Therefore, this trial was blinded to subjects and statisticians only. The statistical analyst was a non-subject and was not aware of the patient's treatment or the trial protocol. For all patients who participated in acupuncture, blinded evaluation questions were asked one week after acupuncture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental): Bilateral Zusanli (ST36) and Sanyinjiao (SP6) acupoints were selected. After obtaining deqi sensation upon needle insertion, an electroacupuncture device was connected to each of the selected acupoints. A sparse-dense wave mode was chosen, with an intensity ranging from 0.5 to 2 mA, adjusted according to patient tolerance. The needles were retained for 20 minutes before removal. The electroacupuncture treatment was initiated on the same day as the commencement of the immunotherapy cycle, administered once daily for a total of five sessions, ensuring that each immunotherapy cycle was synchronized with electroacupuncture treatment. The overall treatment consisted of 4 to 6 cycles.
  Interventions: Other: Electroacupuncture (EA)
- Sham electroacupuncture group (Sham Comparator): Bilateral Zusanli (ST36) and Sanyinjiao (SP6) acupoints were selected. Electroacupuncture devices were connected to these acupoints. A sparse-dense wave mode was utilized, with an intensity ranging from 0.5 to 2 mA, and the needles were retained for 20 minutes before removal. In the sham electroacupuncture group, no manual manipulation was performed. The placement of electrodes and other treatment settings were identical to those in the electroacupuncture group, but without skin penetration, electrical output, or needling techniques to induce deqi. Electroacupuncture treatment was initiated on the same day as the start of the immunotherapy cycle, administered once daily for a total of five sessions, ensuring synchronization with each immunotherapy cycle. The overall treatment regimen consisted of 4 to 6 cycles.
  Interventions: Other: Sham electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture (EA) — In the electroacupuncture group, bilateral Zusanli (ST36) and Sanyinjiao (SP6) points were selected for needling. Upon achieving the "deqi" sensation, the electroacupuncture device was connected to the needles at both points. A dispersed-dense wave was applied with an intensity ranging from 0.5 to 2 mA, adjusted according to the patient's tolerance. The needles were retained for 20 minutes, after which they were removed.
  Arms: Electroacupuncture group
Other: Sham electroacupuncture — In the sham electroacupuncture group, bilateral Zusanli (ST36) and Sanyinjiao (SP6) points were selected for sham electroacupuncture intervention, which did not receive manual manipulation. The electrode placement and other treatment settings were identical to those in the electroacupuncture group, but no skin penetration, electrical output, or needle techniques were applied to induce the sensation of "deqi." No genuine electroacupuncture stimulation was administered in this group.
  Arms: Sham electroacupuncture group

SUMMARY:
The goal of this clinical trial is to elucidate the clinical efficacy and safety of electroacupuncture combined with PD-1 inhibitor therapy in elderly patients with advanced non-small cell lung cancer (NSCLC) through a multicenter, randomized controlled clinical trial. The main question it aims to answer is: the combination of electroacupuncture and PD-1 inhibitor therapy has demonstrated significant improvements in both clinical efficacy and safety profiles among elderly patients with advanced NSCLC. Researchers will compare a sham electroacupuncture group combined with PD-1 inhibitor therapy (serving as the control group) to see if the intervention group exhibits superior therapeutic efficacy and safety outcomes. Participants will be randomly assigned to one of two groups: an electroacupuncture combined with an immune checkpoint inhibitor group, or a sham electroacupuncture combined with an immune checkpoint inhibitor group. The immune checkpoint inhibitor will be administered on a 21-day cycle, with a total of 4 to 6 treatment cycles, followed by the option for maintenance therapy. Electroacupuncture treatment will commence on the same day as the initiation of the immune checkpoint inhibitor cycle, administered once daily for a total of five sessions per cycle, with 4 to 6 cycles in total. The primary outcome measure is progression-free survival (PFS). Secondary outcomes include objective response rate (ORR), quality of life, immune function, traditional Chinese medicine syndrome scores for lung cancer, and safety parameters. This study aims to establish the efficacy and safety of electroacupuncture combined with PD-1 inhibitors in elderly patients with advanced NSCLC. Additionally, peripheral non-coding RNA will be collected at baseline to analyze differentially expressed genes, thereby identifying molecular predictive biomarkers for patients who may benefit most from this combined treatment approach.

DETAILED DESCRIPTION:
This study is designed in accordance with the standards of evidence-based medicine, employing a multicenter, randomized controlled clinical trial framework. It aims to provide high-quality evidence regarding the clinical efficacy of acupuncture combined with PD-1 inhibitors in elderly patients with advanced NSCLC.

Acupuncture has been shown to exert bidirectional regulatory effects on the tumor immune microenvironment. This study seeks to elucidate the predictive biomarkers through which acupuncture synergizes with immune checkpoint inhibitors to improve clinical outcomes in elderly patients with advanced NSCLC. Additionally, it explores the clinical and biological characteristics of the patient population that may derive the greatest benefit from this combined therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IIIB-IV non-small cell lung cancer (NSCLC) confirmed by histopathological or cytological diagnosis.
* Patients with negative driver gene mutations, as determined by genetic testing or other molecular biological methods, to exclude common driver mutations such as EGFR mutations and ALK rearrangements.
* Patients aged ≥65 years, with consideration for the patients' overall physical condition. Additional assessments will be conducted if there are comorbidities or other factors that may affect their physical status.
* PD-L1 tumor proportion score (TPS) ≥1%.
* Estimated survival time >3 months, as determined by clinical evaluation based on the patient's overall condition, tumor progression, and response to treatment.
* ECOG performance status score of 0-2.
* Patients with good treatment compliance, who are willing to sign an informed consent form, indicating their understanding and agreement to adhere to the study protocol for treatment and follow-up.

Exclusion Criteria:

* Patients with a history of or concurrent other malignancies within the past 5 years.
* Patients with severe organ dysfunction or other serious comorbidities, such as heart failure (NYHA Class III-IV), hepatic or renal insufficiency, as assessed by routine examinations including liver function tests, renal function tests, and electrocardiograms.
* Patients with untreated central nervous system metastases. Only those who have undergone at least one course of systemic or surgical treatment and have been confirmed to have stable disease by imaging studies will be included.
* Patients with psychiatric disorders, including a history of severe mental illnesses (e.g., schizophrenia, bipolar disorder) that require pharmacological treatment for control.
* Patients with a history of multiple drug allergies or an allergic constitution, particularly those who have experienced severe allergic reactions such as anaphylactic shock or allergic rashes.
* Patients with active autoimmune diseases or infectious diseases, including but not limited to active or chronic viral hepatitis, active pulmonary tuberculosis, or other infectious or autoimmune conditions deemed by the clinical investigator to potentially affect the study.
* Patients who are pregnant or breastfeeding.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | Defined as the time interval from the date of enrollment to the first documented occurrence of disease progression or death from any cause, whichever comes first. This outcome will be assessed up to 100 months.
  Defined as the interval from the time of enrollment to the first documentation of disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
This decision may stem from concerns regarding privacy or ethical issues associated with data sharing, or because the research data is considered proprietary and not intended for public disclosure.